CLINICAL TRIAL: NCT04804150
Title: Daily Socket Comfort in Transtibial Amputee With an Active Vacuum Suspension System : a Randomized, Multicenter, Double-blind N-of-1 Trial
Brief Title: Daily Socket Comfort in Transtibial Amputee With an Active Vacuum Suspension System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A01309-30
Record Dates: First submitted 2021-03-03; First posted 2021-03-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Amputation
Keywords: Amputation; Elevated vacuum; Prosthetic suspension system; Vacuum-assisted suspension; N-of-1 Trial

STUDY DESIGN:
Intervention Model Description: Multiple N-of-1 trial. : the principle is to evaluate intensively and prospectively a small group of subjects, each case being its own comparator
Masking Description: The medical device will be active (plugged) or inactive (unplugged), but the patient nor the investigator won't know if the medical device is active(plugged) or inactive (unplugged).
  After one-month accommodation period, patient will be randomly distributed into active or inactive vacuum 7 to 28 days phases with at least three phase change and a maximum of 50 days. The randomization will use a phase length ABAB randomization rather than block randomization commonly used in drug trials. However, because the patient has to come to the rehabilitation center at each phase change which would not allow the patient and the assessors to be blind to the next phase content, phases of a duration >14, will be further randomized into two half-phases of the same content with a placebo visit between the two half-phases, in order to keep the blinding. All sequences containing 3 true transition of activation/inactivation of the medical device and up to 3 placebo transitions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medical Device active or inactive (Experimental): The medical device will be active, or inactive. Randomization will define when and how long time the medical device will plugged and active, and when and how long time the medical device will be unplugged and inactive. The patient won't know if the medical device is active or not
  Interventions: Device: Vacuum suspension system active or inactive

INTERVENTIONS:
Device: Vacuum suspension system active or inactive — The device will be plugged in, or won't be plugged in, depending of the randomization. The patient and the investigator will not know whether the device is plugged in or not, and if the medical device is active or not

SUMMARY:
The aim of this study is to evaluate the contribution of the vacuum suspension system in an ecological environment on the fitting's comfort compared to the vacuum suspension system inactive system in a multicenter prospective, randomized, double-blind, multiple N-of-1 trial.

In order to assess the therapeutic effect of the vacuum suspension system, given the heterogeneity of the population and the small number of patients eligible for the study, the multiple N-of-1 trial seems to us to be the methodology. The principle is to evaluate intensively and prospectively a small group of subjects, each case being its own comparator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age.
* Unilateral transtibial amputation for more than 6 months.
* Equipped for more than 3 months with a Seal-in™ liner without the vacuum suspension system.
* Equipped with an ESAR(Energy Storing and Return) foot with the vacuum suspension system
* Patient meeting the criteria of ICF(International Classification of Functioning, Disability and Health) classification d4602 and/or d4608
* Presenting some discomfort in the socket evaluated by a SCS ≤ 7/10
* Absence of severe comorbidity
* Patient with a smartphone and a functional 4G connection

Exclusion Criteria:

* Cognitive impairment that does not allow instructions to be followed
* Have already been equipped with the evaluated vacuum suspension system
* Pregnant women
* Patient subject to a legal protection measure
* Patient not affiliated with social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Confort change assessment | 50 days
  Assess the impact of the vacuum suspension system on the fitting's comfort compared to the vacuum suspension system inactive system with a daily evaluation on Socket Comfort Score [Scale : On a 0 - 10 scale : 0 represents the most uncomfortable socket fit you can imagine, and 10 represents the most comfortable socket fit]

SECONDARY OUTCOMES:
Change in daily wearing time of the prosthesis | Every day during 50 days
  Declarative, in hours
Change in the daily number of steps | Every day during 50 days
  Measured with a pedometer
Assessment of the stump volume variation | Every day during 50 days
  The stump volume variation will be assessed by 2 questions :
  How many times have you removed your prosthesis during the day (not counting the evening's removal) to add compensation sheaths? " 0, 1, 2, 3, 4, >4
  Did you have the fear at one (or more) moment(s) of the day, of losing your prosthesis, that it would come off by itself? " Visual Analogue Scale (VAS) of 0: no not at all at 10 = yes a lot
Assessment of limb-prosthesis coaptation | Every day during 50 days
  The limp-prosthesis coaptation will be assessed by 2 questions :
  "Do you feel that you have mastered your prosthesis, that it is one with you?" VAS from 0 = not at all to 10 =perfectly
  "Do you feel a piston movement of your prosthesis when walking (sensation of vertical movement of the prosthesis in relation to the stump when walking)?" VAS from 0 = not at all to 10 = yes a lot
Change L-Test of Functional Mobility | Up to 50 days
  The L Test is a timed ambulation over 20 meters, which includes two sit to/from stand transfers and three turns
Change in 6 Minute Walk Test (6MWT) | Up to 50 days
  The 6MWT is simply a record of the distance traveled by a given patient at his or her self-selected walking speed over a period of six minutes. All that is required is a stopwatch and a walking corridor or track of known distance. Those administering the test should avoid walking with or in front of test subjects to avoid pacing individuals outside of their self-selected walking speed
Change in patient satisfaction with device: Quebec User Evaluation of Satisfaction with Assistive Technology | Up to 50 days
  Measured with QUEST scale. The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) is a 12-item outcome measure that assesses user satisfaction with two components, Device and Services. Scores of 1 indicate dissatisfaction and scores of 5 indicate high satisfaction
Change in confidence in maintaining balance while doing daily activities | Up to 50 days
  Measured by the simplified Activities-specific Balance Confidence Scale (ABC-S)

CONTACTS AND LOCATIONS:
Overall Officials: REMI KLOTZ, MD, Principal Investigator — LA TOUR DE GASSIES
Locations (3):
- France (3):
  - Clinique de Provence-Bourbonne, Aubagne
  - La Tour de Gassie, Bruges
  - Chu Clermont Ferrand, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Klotz R, Emile G, Daviet JC, De Seze M, Godet J, Urbinelli R, Krasny-Pacini A. Daily socket comfort in transtibial amputee with a vacuum-assisted suspension system: study protocol of a randomized, multicenter, double-blind multiple N-of-1 trial. BMC Sports Sci Med Rehabil. 2023 Jul 14;15(1):85. doi: 10.1186/s13102-023-00694-4. PMID 37452356